CLINICAL TRIAL: NCT07253506
Title: Turkish Adaptation, Validity, and Reliability Study of the Patient Experience With Treatment and Self-Management Scale in Stroke Patients
Brief Title: Turkish Adaptation, Validity, and Reliability Study of the Patient Experience With Treatment and Self-Management Scale in Stroke
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: istftrrr
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study will include individuals aged 18-80 years who have been clinically diagnosed with stroke and have spent at least one month at home after discharge. Sociodemographic and clinical characteristics will be recorded. Functional status will be assessed using the Modified Rankin Scale, Brunnstrom Stages, and the Modified Barthel Index. Ambulation status will be documented with the Holden Scale.

The scale will first be translated into Turkish and then back-translated into English by a bilingual expert whose native language is English. The Turkish version of the scale will be administered to patients. Two independent evaluators will apply the scale twice, one week apart.

Validity will be examined by analyzing the relationship between the scale and the Stroke Impact Scale and the Treatment Burden Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke (ischemic or hemorrhagic).
* Having spent at least 1 month at home after hospital discharge (to capture post-acute home care/rehabilitation burden).
* Community-dwelling individuals aged 18-80 years.
* Adequate Turkish reading-writing and communication ability.
* Ability to provide informed consent.
* In cases of mild aphasia, ability to complete the questionnaire independently or with support.

Exclusion Criteria:

* History of subarachnoid hemorrhage.
* Inability to communicate effectively due to severe aphasia or severe cognitive impairment.
* Terminal illness (life expectancy < 6 months).
* Inability to complete the questionnaire reliably due to a psychiatric disorder.
* Acute phase (those hospitalized or before discharge).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical diagnosis of stroke (ischemic or hemorrhagic).
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
PETS-Stroke scale | Baseline
  The primary measure, the PETS-Stroke scale, evaluates patients' experiences with treatment and self-management; its scoring system is based on subscale scores typically transformed to 0-100, with higher values reflecting greater perceived burden or difficulty in treatment and self-management.

SECONDARY OUTCOMES:
The Modified Rankin Scale | Baseline
  The Modified Rankin Scale will be used to assess overall functional status; this scale measures global disability on a 0-6 range, with higher scores indicating greater dependence.
Modified Barthel Index | Baseline
  Independence in activities of daily living will be assessed with the Modified Barthel Index, scored between 0 and 100, where higher scores reflect greater functional independence.
Stroke Impact Scale | Baseline
  To assess construct validity, the Stroke Impact Scale will be used; it measures the impact of stroke on domains such as daily activities, mobility, hand function, communication, emotion, memory, and participation, with domain scores transformed to a 0-100 scale in which higher scores represent better status.
Treatment Burden Questionnaire | Baseline
  Treatment burden will be evaluated with the Treatment Burden Questionnaire, where items are scored from 0 to 10, and higher scores indicate greater perceived treatment burden.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)